CLINICAL TRIAL: NCT04800757
Title: VALES+Tú: Targeting Psychosocial Stressors to Reduce Latino Day Laborers Injury Disparities
Brief Title: VALES+Tú: Targeting Psychosocial Stressors to Reduce Latino Day Laborers (LDL) Injury Disparities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Maria Eugenia Fernandez-Esquer, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-18-0337; 1R01MD012928 (NIH)
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Work-related Injury
Keywords: latino day laborers
MeSH Terms: interventions — Population Groups; Standard of Care

STUDY DESIGN:
Intervention Model Description: Cluster randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- individual (Brief Motivational Intervention) (Experimental)
  Interventions: Behavioral: individual -Brief Motivational Intervention (BMI)
- Group (Group Problem Solving) (Experimental)
  Interventions: Behavioral: Group (Group Problem Solving)
- Standard of Care (Placebo Comparator)
  Interventions: Behavioral: Standard of Care (OSHA 10 Safety Cards)

INTERVENTIONS:
Behavioral: individual -Brief Motivational Intervention (BMI) — A baseline survey will be administered prior to the session.Sessions will be initiated by exploring working conditions and psychosocial factors that may influence risk for work related injuries. If the LDL is motivated to change the target behavior, a 'change plan' will be developed which involves identifying reasons for change, goals in making change, specific actions and timelines, and others who may help the person change. The final step will be the development of a personal safety plan to reduce work place risks and a discussion of the following topics: (a) how they will know if their plan is successful, (b) potential obstacles, and (c) what the worker can do if the plan does not work. Finally,each worker will be asked to write and sign a personal pledge ("Mi Promesa") to implement his own safety plan.Follow-up surveys will be conducted 4 weeks after the baseline survey.
  Arms: individual (Brief Motivational Intervention)
Behavioral: Group (Group Problem Solving) — Participants will be administered a baseline survey prior to session. The GPS intervention consists of a discussion between 2-5 LDLs and a trained group facilitator. The sessions will last 30-45 minutes and are intended to encourage and support Latino day laborers (LDL) to act to reduce work-related hazards and promote worksite safety. The intervention combines four participatory and group problem solving activities to engage in collaborative learning: an icebreaker, the risk identification, action planning, and Nuestra Promesa (Our Pledge). The last activity requires LDL to select a risk reduction behavior and then to fill out and sign a card detailing a pledge to implement a safety plan. Follow up surveys will be conducted four weeks post intervention, to assess participants' change in attitudes, beliefs, and risk reducing behavior and their implementation or their safety plan.
  Arms: Group (Group Problem Solving)
Behavioral: Standard of Care (OSHA 10 Safety Cards) — Participant will be administered a baseline survey prior to the session.Participants in this standard of care control group will receive four wallet size cards with information about risk reduction strategies to deal with the four hazards responsible for most workplace fatalities in Texas: falls, struck by, heat exposure and cuts. The laminated cards are adapted from OSHA's website publicly available materials in Spanish for workers with limited literacy.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to determine the efficacy of VALES+Tú in reducing hazardous exposures at work and to determine the mediating effect of psychosocial stressors on VALES+Tú primary outcomes

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Hispanic or Latino
* be present at the corner for the purpose of looking for work

Exclusion Criteria:

* have not been previously hired to work at a corner
* symptoms of COVID-19 in the previous 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Eugenia Fernandez-Esquer, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: corners
Groups:
- Group (Group Problem Solving): Group (Group Problem Solving): Participants will be administered a baseline survey prior to the session. The group problem solving intervention will consist of a discussion between 2-5 LDLs and a lay health promoter trained as a group facilitator. The sessions are expected to last 30-45 minutes and are intended to encourage and support Latino day laborers (LDL) to take action to reduce work-related hazards and promote worksite safety for themselves and their co-workers. The intervention combines four participatory and group problem solving activities to engage in collaborative learning: an icebreaker, the risk identification, action planning, and Nuestra Promesa (Our Pledge). The last activity requires each LDL to select a risk reduction behavior and then to fill out and sign a card detailing a pledge to implement a safety plan. Follow up surveys will be conducted over the phone, four weeks post intervention, to assess participants' change in attitudes, beliefs, and risk reducing behavior and their implementation or their safety plan.
Period: Overall Study
Arm/Group | Standard of Care | Individual (Brief Motivational Intervention) | Group (Group Problem Solving)
Started | 113; 10 corners | 102; 10 corners | 110; 10 corners
Completed Baseline Assessment | 112; 10 corners (One subject did not complete baseline survey) | 100; 10 corners (2 subjects did not complete baseline survey) | 106; 10 corners (4 subjects did not complete baseline survey)
Completed Post-Intervention Assessment | 91; 10 corners | 82; 10 corners | 75; 10 corners
Completed | 91; 10 corners | 82; 10 corners | 75; 10 corners
Not Completed | 22; 0 corners | 20; 0 corners | 35; 0 corners

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for the 318 participants who completed the baseline assessment. Age was not collected for one participant in the BMI arm.
Groups:
- Group (Group Problem Solving): Group (Group Problem Solving): Participant will be administered a baseline survey prior to the session.The group activity intervention will consist of a discussion between 3-4 LDL and a promotor (a peer LDL) trained as a group facilitator. The sessions are expected to last 20-30 minutes and are intended to provide an opportunity for the participants to work on a safety problem together, get to know each other, and enhance their mutual safety through mutual support.Follow-up surveys will be conducted 4 weeks after the baseline survey. Oral informed consent will be obtained prior to each follow-up survey. The follow-up surveys will reassess participants' work and injury experiences and experiences with the safety intervention they were provided - safety cards, change plan, or safety plan.
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Individual (Brief Motivational Intervention) | Group (Group Problem Solving) | Total
Number analyzed (Participants) | 112 | 100 | 106 | 318
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was not collected for one participant in the BMI arm.
  years
    number analyzed (Participants) | 112 | 99 | 106 | 317
    (all) | 46 (12.3) | 44.1 (11.3) | 46.5 (11.3) | 45.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 112 | 100 | 106 | 318
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 112 | 100 | 106 | 318
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 112 | 100 | 106 | 318
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 112 | 100 | 106 | 318

OUTCOME MEASURES:

1. Primary Outcome: Change in Work Hazard Exposure as Assessed by a Survey
Description: Total score on the work hazard exposure survey ranges from 1 - 4, with a higher score indicating greater work hazard exposures. The data are reported as score at post-intervention minus score at baseline.
Time Frame: Baseline, 4 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care | Individual (Brief Motivational Intervention) | Group (Group Problem Solving)
Number analyzed (Participants) | 91 | 82 | 75
score on a scale | -0.25 (0.56) | -0.07 (0.52) | -0.26 (0.50)

2. Primary Outcome: Change in Work Conditions as Assessed by a Survey
Description: Total score on the work conditions survey ranges from 1 - 4, with a higher score indicating greater adverse work conditions. The data are reported as score at post-intervention minus score at baseline.
Time Frame: Baseline, 4 weeks post intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Standard of Care | Individual (Brief Motivational Intervention) | Group (Group Problem Solving)
Number analyzed (Participants) | 91 | 82 | 75
score on a scale | -0.21 (0.54) | -0.21 (0.49) | -0.38 (0.59)

3. Secondary Outcome: Change in Safety Practices as Assessed by a Survey
Description: The score for each of the 22 safety practices items ranged from 1-4, with a higher score indicating greater safety practice. The total score for the complete scale consisting of all 22 items is the average of items responded to and also ranged from 1-4. Separate scores for each subscale were computed similarly. The first subscale consisted of eight items; the second consisted of four items, and the third consisted of three items--the score for each subscale ranged from 1-4, with a higher score indicating greater safety practice. There were seven original items that were not associated with the subscales derived from the factor analyses. The data are reported as scores at post-intervention minus scores at baseline.
Time Frame: Baseline, 4 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard of Care | Individual (Brief Motivational Intervention) | Group (Group Problem Solving)
Number analyzed (Participants) | 91 | 82 | 75
score on a scale
  Safety Practices: All Items | -0.11 (0.49) | 0.03 (0.59) | 0.03 (0.53)
  Safety Practices: Preparation Safety | -0.15 (0.71) | 0.01 (0.80) | 0.01 (0.73)
  Safety Practices: Harm Mitigation | 0.02 (0.61) | -0.01 (0.59) | 0.06 (0.64)
  Safety Practices: Proactive Communication | -0.16 (0.93) | 0.04 (1.13) | 0.10 (0.90)

4. Secondary Outcome: Number of Participants That Implemented the Safety Plan as Assessed by a Survey
Description: Participants were asked if they implemented the safety plan and they were asked to answer as yes, no or partially
Time Frame: 4 weeks post intervention
Population: The participants in the standard of care arm did not make a safety plan; therefore, safety plan data were not collected for the standard of care arm. Also, data for this outcome measure were not collected from 34/82 participants in the Brief Motivational Intervention arm and 34/75 participants in the Group Problem Solving arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Individual (Brief Motivational Intervention) | Group (Group Problem Solving)
Number analyzed (Participants) | 0 | 48 | 41
Participants
  No | 0 | 5 | 5
  Yes | 0 | 18 | 24
  Partially | 0 | 25 | 12

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Standard of Care | Individual (Brief Motivational Intervention) | Group (Group Problem Solving)
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/100 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/100 | 0/106
Other Adverse Events (participants affected / at risk) | 0/112 | 0/100 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT04800757/Prot_SAP_000.pdf